CLINICAL TRIAL: NCT04807023
Title: Decompensation of Cirrhosis and Iron Metabolism
Acronym: DeCiFer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC20_8895_DeCiFer; 2020-A02454-35 (Other: N° IDRCB)
Record Dates: First submitted 2021-03-16; First posted 2021-03-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-03

CONDITIONS: Cirrhosis
Keywords: Decompensation of cirrhosis; Iron metabolism
MeSH Terms: conditions — Fibrosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: blood sampling — blood sampling

SUMMARY:
Iron is a crucial metal whose metabolism is tightly regulated. Iron deficiency or iron overload are both deleterious at the cellular, organic and systemic levels. In line with the major role of the liver in iron homeostasis, links between iron metabolism and acute on chronic liver failure have been highlighted. Nevertheless, due to the difficulty of accurately assessing iron metabolism in this situation, therapeutic intervention on iron metabolism in this setting is currently not codified.

A better understanding of these mechanisms is therefore essential, in particular by characterizing the impact of exposure to non-transferrin-bound iron in acute on chronic liver failure on short-term mortality.

Overall, a better understanding of the physiopathological mechanisms of iron should allow to optimize the martial balance in this condition and also improve therapeutic approaches.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Diagnosis of cirrhosis, previously known or not, of any etiology, histologically proven or not.
* Hospitalization for acute on chronic liver failure:
* Ascites decompensation.
* Or spontaneous infection of the ascites fluid (defined as PNN > 250/mm3 of ascites).
* Or digestive hemorrhage related to portal hypertension (digestive fibroscopy showing active bleeding or stigmas of recent bleeding from esophageal and/or gastric varices).
* Or hepatic encephalopathy (clinically defined +/- increase in ammonia and/or by electroencephalogram and classified in stages according to West-Haven).
* Or hepato-renal syndrome (HRS-AKI criteria, EASL 2018).
* Or bacterial infection (defined by a bacteremia identified by at least one blood culture and/or an infectious site authenticated on imaging).
* Or Acute Alcoholic Hepatitis (histologically proven or not).
* Non-opposition of the patient, relative or legal representative.

Exclusion Criteria:

* Treatment with oral or intravenous iron in the month prior to hospitalization.
* Implementation of a TIPS in the month prior to admission.
* Presence of hepatocellular carcinoma with an expected survival < 3 months or any other progressive cancer.
* Adult person subject to legal protection (safeguard of justice, curatorship, guardianship), person deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with diagnosis of cirrhosis hospitalized for acute on chronic liver failure
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-05-17 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Mortality | day 28

SECONDARY OUTCOMES:
Serum levels of abnormal iron | days 0, 2, 7 and 14
Ceruloplasmin ferroxidase activity | days 0, 2, 7 and 14
hepcidin blood levels | days 0, 2, 7 and 14
Ferritinemia | days 0, 2, 7 and 14
transferrinemia | days 0, 2, 7 and 14
transferrin saturation coefficient | days 0, 2, 7 and 14
Blood levels of manganese | days 0, 2, 7 and 14
Occurrence of complications | during hospitalization and a maximum of 28 days after admission
Bacterial infection | during hospitalization and a maximum of 28 days after admission
fungal infection | during hospitalization and a maximum of 28 days after admission

CONTACTS AND LOCATIONS:
Overall Officials: Giguet Baptiste, Principal Investigator — CHU Rennes
Locations (1):
- CHU Rennes, Rennes, France